CLINICAL TRIAL: NCT04138134
Title: Impact of Reactivation of Autophagy Through Spermidine on Venous Endothelial Function
Brief Title: Autophagy and Venous Endothelial Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: Principal investigator: Giacomo Frati (Unknown); Co-investigator: Francesco Pompeo (Unknown)
Responsible Party: Principal Investigator, Maurizio Forte, Principal investigator, Neuromed IRCCS
Other Study IDs: 9-2019
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Venous Disease
Keywords: autophagy; spermidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients subjected to saphenectomy due to chronic venous insufficiency or varicose veins
- Group 2: Patients with atherosclerotic obstructive disease of lower limbs

SUMMARY:
The molecular mechanisms involved in venous endothelial dysfunction are largely unknowns. Autophagy is an intracellular mechanism devoted to the removal of damaged cytoplasmic elements. Previous evidence demonstrated that activation of autophagy exerts beneficial effects in the cardiovascular system, reducing cardiac damage and improving cardiac function in response to stress. However, the association between venous endothelial dysfunction and autophagy remains to be characterized. In this study the investigators will test whether reactivation of autophagy through a natural compound (spermidine) is able to improve vascular function in saphenous veins derived from patients subjected to saphenectomy. The same outcome will be evaluated in saphenous veins isolated from patients with atherosclerotic obstructive disease of the lower limbs subjected revascularization through implantation of venous by-pass.

DETAILED DESCRIPTION:
Endothelial dysfunction contributes to different cardiovascular diseases, such as atherosclerosis, myocardial infarction, stroke and peripheral artery diseases. Recent evidence also demonstrated that endothelial dysfunction is associated with vascular venous diseases. In this regard, venous endothelial dysfunction contributes to the development of varicose veins and deep vein thrombosis. Disequilibrium in endothelial function is also present in venous traits derived from saphenous veins which are routinely used as aortocoronary by-pass. The molecular mechanisms involved in venous diseases require further investigations. Autophagy, the intracellular mechanism devoted to the removal of dysfunctional or senescent cytoplasmic elements may represent a new therapeutic target for the treatment of vascular diseases. In this regard, it has been demonstrated that the enhancement of autophagy limits cardiac injury in pre-clinical models of cardiovascular diseases. However, the association between autophagy and vascular disease is still unknown in humans. Spermidine is a natural activator of autophagy which has been demonstrated to extend lifespan in mice and to reduce cardiac dysfunction through autophagy-dependent mechanisms. The objectives of this study will be the following: 1) to test whether spermidine is able to improve vascular function and to reduce oxidative stress in saphenous veins obtained from patients subjected to saphenectomy due to chronic venous insufficiency or varicose veins; 2) to test whether spermidine is able to improve vascular function in saphenous veins derived from patients with atherosclerotic obstructive disease of lower limbs subjected to revascularization through implantation of arteriosus by-pass. In a different set of experiments, the investigators will also test whether vein portions incubated with spermidine show increased autophagy and decreased markers of oxidative stress with respect to controls. The investigators expect that venous segments treated with spermidine will show an amelioration of endothelial function

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects undergoing saphenectomy
* Patients with chronic venous insufficiency
* Patients with varicose veins
* Eligible subjects undergoing peripheral artery revascularization through implantation of venous by-pass derived from saphenous vein
* Acceptance and signature of the informed consent

Exclusion Criteria:

* Chronic and acute Inflammatory diseases
* Immunological and rheumatic diseases
* Pre-existing or ongoing neoplasms
* Infectious diseases
* Previous organ transplantation
* Treatment with pharmacological therapies able to modulate autophagy, i. e. rapamycin and derivative compounds (rapalogues).
* Antioxidant therapies in the last three months
* Patients with surgical technical complications

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Subjects affected by chronic venous insufficiency or varicose veins undergoing surgical procedure of saphenectomy.
  * Patients with atherosclerotic obstructive disease of the lower limbs subjected revascularization through implantation of venous by-pass.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of endothelial function in venous samples from patients with venous insufficiency before and after treatment with autophagy enhancer spermidine | Immediately after the sampling
  Ex vivo vascular reactivity experiments performed on isolated veins treated or not with spermidine ex vivo.

SECONDARY OUTCOMES:
Impact of autophagy on endothelial venous function | 6 months
  Quantification by immunoblot of markers of autophagy (LC3, p62, Beclin1, Atg5, Atg7, Ulk1) and its statistical correlation with venous endothelial function
Correlation between autophagy, oxidative stress and endothelial function | 6 months
  Quantification by immunoblot of markers of autophagy and oxidative stress and statistical correlation with venous endothelial function

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy